CLINICAL TRIAL: NCT06190132
Title: Omega-3 Fatty Acids Versus Gabapentin in Uremic Pruritus in Hemodialysis Patients.
Brief Title: The Effect of Omega-3 Fatty Acids Versus Gabapentin in Uremic Pruritus in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 768/2022
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-10

CONDITIONS: Uremic Pruritus in Hemodialysis Patients
Keywords: Hemodialysis patients
MeSH Terms: interventions — Fatty Acids, Omega-3; Gabapentin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A allocated to treatment with omega 3 fatty acids for 4 weeks then after 6 weeks washout period, the patients received gabapentin for 4 weeks
  Interventions: Drug: Omega 3 fatty acid, gabapentin
- Group B (Active Comparator): Group B allocated to treatment with gabapentin for 4 weeks then after 6 weeks washout period, the patients received omega 3 fatty acids for 4 weeks
  Interventions: Drug: Omega 3 fatty acid, gabapentin

INTERVENTIONS:
Drug: Omega 3 fatty acid, gabapentin — To study the effect of omega 3 fatty acids on uremic pruritus in prevalent hemodialysis patients versus the effect of gabapentin
  Other Names: Gabapentin

SUMMARY:
omega-3 fatty acids versus gabapentin in uremic pruritus in hemodialysis patients.

DETAILED DESCRIPTION:
Patients who were enrolled in the study used no antipruritic therapy for at least 2 weeks before the study. The patients were randomly assigned to Group A, or Group B. Patients in Group A (25participants) were allocated to treatment with omega-3 daily (2capsules of 1gm omega-3 a day) (Shayanpour et al.,2019). Patients in Group B (25 participants) received gabapentin (one capsule of gaptin 100mg thrice weekly post HD session) (KDIGO Clinical practice guidelines,2019) Patients in the 2 groups received treatment for four weeks then after washout period(6 weeks), the treatment was changed between the 2 groups. pruritus severity was assessed by 5D-Itch score before the study and at the end of each treatment period. Throughout the study, the level of PGE2 and the pruritus severity was measured at the baseline before treatment, after 4 weeks and after 14 weeks (post treatment) by 5-D itch scale.

5-D itch scale was made to be used for outcome measurement in clinical trials. It depends on five main domains for measurement of pruritus severity which are (duration, degree, direction, disability and distribution) (Elman et al.,2010). The score of each domain is made separately then the scores of all domains summed together to obtain the total 5-D score pruritus). Patients with score 5 or less considered having no itching and patients with scores from 6 to 25 considered itch patients.

The total 5-D score can be classified into:

1. The score of 6-10 is considered mild pruritus.
2. The score of 11-20 is considered moderate pruritus.
3. The score of 21-25 is considered severe pruritus.

So the study group will fulfill the following criteria :

1. According to 5D itch score a total score of 6-25 points
2. Meet the international diagnostic criteria for uremic pruritus.
3. Meet the exclusion criteria of the study. The total score can range from 5(which mean no pruritus) to 25 (which mean most severe

ELIGIBILITY:
Inclusion Criteria: prevalent hemodialysis patients >18 years undergoing dialysis who are co operative and not receiving topical or systemic treatment for uremic pruritus for at least 2 week patients who meet the international diagnostic criteria for uremic pruritus

Exclusion Criteria:

Patients with primary dermatological disease causing itching as atopic dermatitis, psoriasis, scabies, drug reaction Patients with any systemic disease that can cause pruritus as hepatic cholestasis , active infections (hepatitis B, and hepatitis c PCR positive, HIV) Patients under steroid treatment. current treatment of uremic pruritus. Concomitant malignancy (Hodgkins lymphoma, leukemia, multiple myeloma) Kidney transplantation (immunosuppressive medications Contraindications to omega 3 as patients using anticoagulants, or patients who have bleeding tendency, chronic diarrhea, history of malabsorption or allergic reaction to omega 3 Contraindications to gabapentin as in patients who have depression , suicidal thoughts, myasthenia Gravis, skeletal muscles disorder, patients who have history of allergic reactions to gabapentin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
5 Dimensions itch scale, prostaglandin E2 | 14 weeks
  5 Dimensions itch scale used for measurement of pruritus severity and outcome measurement in clinical trials score from 6 to 25 considered to have pruritus, PGE2 used for assessment of pruritus as its produced in cases of inflammation, involved in pain sensation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt